CLINICAL TRIAL: NCT01551251
Title: Tumor-Associated Macrophages Correlate With Response and Outcomes in Advanced Non-Small Cell Lung Cancer After First Line Treatment.
Brief Title: Tumor Associated Macrophage in Advanced Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: 100-0522B
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2011-04

CONDITIONS: Advanced Nonsmall Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — All specimens were fixed in 10% buffered formalin and embedded in paraffin according to standard procedures. All of the tissues were fixed immediately after biopsy, with time from tissue acquisition to fixation as short as possible. Serial sections (4 μm thickness) placed on positively charged slides (Menzel-Glasser, German) were used for immuno-histochemistry.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Advanced NSCLC with high TAM: All patients with advanced non-small cell lung cancer who had been treated at the Linkou Branch of Chang Gung Memorial Hospital were included. Tumor specimens with high TAM were included as one cohort group.
- Advanced NSCLC with low TAM: All patients with advanced non-small cell lung cancer who had been treated at the Linkou Branch of Chang Gung Memorial Hospital were included. Tumor specimens with low TAM were included as one cohort group.

SUMMARY:
The purpose of this study is to investigate the effects of tumor associated macrophage (TAM) in advanced non-small cell lung cancer (NSCLC) patients on the treatment response and outcome of these subjects. Pathologic specimens from tissue bank will be stained by immunostaining methods with CD68 antibody. The clinical treatment response and outcomes will be analyzed between high or low TAM.

ELIGIBILITY:
Inclusion Criteria:

* advanced NSCLC,
* more than 20 years old,
* measurable tumor,
* response and outcome recorded after the first line treatment.

Exclusion Criteria:

* Early stage NSCLC,
* less than 20 years,
* pregnancy,
* unmeasurable NSCLC.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with advanced non-small cell lung cancer (stage IIIb and IV NSCLC) who had been treated at the Linkou Branch of Chang Gung Memorial Hospital between 2006 and 2009 were included.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Response to treatment of advanced NSCLC with high or low TAM. | 2-3 months
  All patients with advanced non-small cell lung cancer (NSCLC) who had been treated were included. The decision of advanced NSCLC treatment was a consensus by the patient and clinician, and approved by team conference (including the oncologists, pulmonologists, pathologists, radiologists, surgeons, radiation oncologists, and nuclear medicine specialists). The tumor response was evaluated using computerized tomography according to the Response Evaluation Criteria in Solid Tumors (RECIST). The treatment response of advanced between high and low TAM patients were compared.

SECONDARY OUTCOMES:
Outcomes of advanced NSCLC with high and low TAM. | 12-24 months
  The outcomes of advanced NSCLC with high and low TAM will be compared. The outcomes include overall survival (OS) and progression-free survival (PFS). Survival curves were estimated by the Kaplan-Meier method while the log-rank test was used to compare the patient survival times per groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tsai Chung, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Taipei, Taipei
  - Sant Paul Hospital, Taoyuan District

REFERENCES:
- [Background] Chen JJ, Lin YC, Yao PL, Yuan A, Chen HY, Shun CT, Tsai MF, Chen CH, Yang PC. Tumor-associated macrophages: the double-edged sword in cancer progression. J Clin Oncol. 2005 Feb 10;23(5):953-64. doi: 10.1200/JCO.2005.12.172. Epub 2004 Dec 14. PMID 15598976